CLINICAL TRIAL: NCT06370637
Title: Comparison of an Enhanced Barrier Cream to Standard of Care for the Treatment of Moisture Associated Skin Damage From Fecal Incontinence in an Ambulatory Population
Brief Title: Testing a Novel Barrier Cream for Fecal Incontinence in an Ambulatory Population
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Scotiaderm (Other)
Collaborators: University of Calgary Cumming School of Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-DRM-004
Record Dates: First submitted 2024-02-13; First posted 2024-04-17 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Moisture Associated Skin Damage; Fecal Incontinence; Incontinence Associated Dermatitis
Keywords: MASD; Moisture Associated Skin Damage; IAD; Incontinence Associated Dermatitis; Fecal Incontinence; Dermategrity; Barrier Cream
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Intervention Model Description: This is a single center, randomized, double-blind, controlled study. This study will follow 40 patients from the wound clinic at the University of Calgary who present with IAD from diarrhea and/or fecal incontinence. Randomizations will be performed at a 1:1 ratio, with 20 patients randomized to the control arm, and 20 patients randomized to the intervention arm.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomizations will be assigned by placing an equal number of control and intervention assignments into opaque envelopes. When a patient is enrolled, the research coordinator will draw an envelope, and the assignment in that envelope will be given to that patient. This process will be repeated for all patients enrolled. Patients will be enrolled until 20 patients are recruited in each study arm. The research coordinator will have a list of the randomizations; this will not be shared with the investigator, the care team, or the participants. Study product will be provided in identical, plain white tubes with labels of arm 1 (control) and arm 2 (intervention). The study coordinator will ensure that participants receive the correct product for their randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Patients randomized to the control arm will be treated with a 15% zinc oxide barrier cream, which is standard of care for MASD.
  Interventions: Other: Barrier Cream
- Investigational Product (Experimental): Patients randomized to the intervention arm will be treated with Dermategrity Everyday Barrier Cream.
  Interventions: Other: Dermategrity Everyday Barrier Cream

INTERVENTIONS:
Other: Barrier Cream — Patients in the control arm will be treated with a 15% zinc oxide barrier cream. Scotiaderm will supply the control product, such that the formula is identical to the intervention with the only difference being the addition of plant extract in the investigational product.
  Arms: Control
Other: Dermategrity Everyday Barrier Cream — Patients randomized to the intervention arm will receive treatment with Scotiaderm's proprietary barrier cream formula. This product contains soy extract for enhanced healing of MASD secondary to fecal incontinence.
  Arms: Investigational Product

SUMMARY:
Liquid stool and diarrhea are associated with an increased risk for moisture-associated skin damage (MASD), and clinical evidence suggests that exposure to liquid stool is associated with severe MASD and extensive erosion of affected skin. There are no known products on the market that treat fecal incontinence or MASD caused by fecal enzyme activity.

Scotiaderm has invented a novel barrier cream (Dermategrity Everyday Barrier Cream) with an enhanced formula containing zinc oxide and soybean extract that inhibits fecal enzymes to protect the skin while preventing further breakdown. Dermategrity Everyday Barrier Cream has shown superior outcomes in comparison to zinc oxide alone in simulated laboratory testing, and promising results have been obtained in clinical case studies. To date, however, there has been no formal clinical testing of this new barrier product in comparison to standard zinc oxide creams.

The purpose of this study is to perform a randomized, controlled clinical study comparing Dermategrity Everyday Barrier Cream to zinc oxide barrier cream to determine if there is a difference in healing, clinical outcomes, and the speed of resolution of MASD symptoms between groups, in an ambulatory patient population.

DETAILED DESCRIPTION:
Moisture associated skin damage (MASD) is a grouping of painful, irritating rashes which occur when a patient has repeated or prolonged exposure to moisture from perspiration, urine and/or feces. Commonly encountered rashes in this group include incontinence-associated dermatitis (IAD) and intertrigo (ITD). These conditions can affect as many as one in five hospitalized patients and up to 50% of intensive care unit patients, putting them at risk of skin breakdown, serious infection, and the development of pressure ulcers. MASD is a common but overlooked and under-reported skin care problem, and there are many gaps in the knowledge of how best to treat these rashes.

Liquid stool and diarrhea are associated with an increased risk for MASD when fecal materials remain in contact with the skin for a prolonged period. Diarrhea is associated with an increased likelihood of IAD in children, and clinical evidence suggests that exposure to liquid stool is associated with severe MASD and extensive erosion of affected skin. Liquid stool is also rich with coliform bacteria, and the gastrointestinal tract acts as a reservoir for various fungal species including Candida, which commonly complicates IAD. Liquid stool contains higher concentrations of proteolytic enzymes with the potential to impair the moisturizing effects of proteins such as filaggrin, and the softening effects of the intrinsic lipids in the skin, both of which are vital in maintaining the barrier functions in skin. These effects are exacerbated by a more alkaline pH and the higher concentrations of active fecal enzymes associated with diarrhea. Research on incontinent patients in the intensive care unit shows that the mean time to development of MASD is 4 days. The presence of liquid stool is an independent risk factor for the development of IAD, with patients developing IAD at a rate of 1.5x that of patients who are continent.

The current standard of care for the treatment and prevention of MASD involves a structured skin care regiment that involves cleansing of the skin to remove excessive moisture and irritants with a pH balanced cleanser, moisturizing the skin when indicated and applying a protective productive product when repeated exposure to moisture is anticipated. There are many factors that influence the choice of moisturizers and protective products, however a Cochrane review of IAD in 2016 noted that there was no evidence that one product was superior to another. Currently, a single-step intervention using disposable washcloths that incorporate cleansing, protecting, and skin restoring agents into a single product (3-in-1 wipes) is widely practiced and helps to maximize adherence to best practices in the treatment and prevention of MASD.

Research has shown that a family of enzyme inhibitors can be isolated from a subset of plants. These plant-based inhibitor peptides (PBIPs) have been well characterized and have been shown to reduce the proteolytic activities of enzymes commonly seen in the digestive tract and feces. PBIPs have demonstrated anticarcinogenic activity against tumor cells in vitro, in animal models, and in human phase II clinical trials. PBIP Concentrates (PBIPCs) have the same anticarcinogenic profile as purified PBIPs and have been developed for human trials. Both PBIPs and PBIPCs are nontoxic, and safety has been reported in numerous clinical studies. Topical PBIPCs have been used safely in clinical studies as hair growth suppressant and to treat skin pigmentation.

Scotiaderm Inc. has developed Dermategrity Everyday Barrier Cream; a topical formulation of a barrier cream containing zinc oxide with PBIPCs from soybeans to be used in the treatment of MASD caused by diarrhea and/or fecal incontinence. The purpose of the proposed research is to evaluate the safety, efficacy, and patient satisfaction with Dermategrity Everyday Barrier Cream for the treatment of Moisture Associated Skin Damage (MASD) caused by fecal incontinence in an outpatient setting. The study design will compare a standard barrier cream for MASD (15% zinc oxide barrier cream) to Scotiaderm's proprietary formula (3% soybean extract in 15% zinc oxide barrier cream) to determine if the plant-based extract enhances the efficacy of treatment.

This is a single center, randomized, double-blind, controlled study. This study will follow 40 patients from the wound clinic at the University of Calgary who present with IAD from diarrhea and/or fecal incontinence. The primary outcomes are the change in erythema score and the patient severity of symptoms score on the GLOBIAD, and patient-reported symptoms on a VAS scale from baseline to days seven and fourteen of treatment. Secondary outcomes will be product-related adverse events, patient-reported satisfaction with the product, and patient-reported healing.

Patients will be followed for two weeks, with a baseline/enrollment visit and follow-up visits occurring on day seven and day fourteen. Both the clinical care team and the patients will be blinded to their group assignment. The research coordinator will provide the clinical team with a plain tube of barrier cream and an envelope outlining the treatment protocol for the study arm the patient has been assigned. The study product will be shipped with the product labels included and these labels will be kept on file by the study coordinator for reference as needed. For all applications the patient (or their personal care aid) will apply the treatment themselves, with instructions provided to patients at the baseline visit.

Between study visits, patients will complete a daily symptoms journal with three VAS questions for pain, itching and burning, record the number of bowel movements/day, as well as note any other relevant symptoms or comments regarding their assigned treatment or their MASD. On days seven and fourteen, patients will present to the clinic for an assessment from the investigator on the status of their rash, which will include completion of the Global IAD Assessment and a VAS Erythema score. Any adverse events or unexpected side effects experienced by the participant will be recorded by the research team during clinic visits and reviewed by the investigator. Patients are instructed to contact the research team immediately if they experience any serious health issues during use of the study product.

Participants will be asked to complete the daily symptom journal for two weeks while participating in the study, and to bring the journal with them to their follow-up visits. For any days that patients report less than 2 applications of the cream, they will be asked to explain why the minimum dosage was not met. On their final visit on day fourteen, patients will return their journal to the study team, and the final clinical assessment will be completed. Patients will be asked to fill out a questionnaire on their satisfaction with the cream used and their opinion on how effective it was at relieving symptoms and treating their rash. Patients will be unblinded once all study activities have been completed.

The primary analysis will focus on the patient severity of symptoms from the Global IAD, the Erythema score, and the patient-reported VAS scores. A repeated measures ANOVA will be used to compare outcomes across time points for each of the independent variables. Efficacy will be assessed by quantifying the change in VAS scores from day 0 to day 7 and day 14. Safety will be assessed by documenting any adverse events/reactions that occur to patients participating in this study. Patient satisfaction with the product will be captured via a standard questionnaire at the conclusion of the study.

It is hypothesized that Dermategrity Everyday Barrier Cream containing will demonstrate an excellent patient-reported safety profile and higher reported rate of healing of MASD due to diarrhea and/or fecal incontinence compared to the standard of care over a two-week period. Furthermore, it is hypothesized that patients will have high satisfaction with the study product.

ELIGIBILITY:
Inclusion Criteria

* ≥18 years of age
* Clinical diagnosis of incontinence-associated dermatitis resulting from diarrhea and/or fecal incontinence.
* Able to provide written informed consent
* Either able to self-administer barrier cream to the affected region OR administer with the assistance of a caregiver

Exclusion Criteria

* History of complex skin disorders (such as psoriasis or eczema)
* Known allergy to any of the ingredients in the study product
* Visual evidence of a bacterial skin infection
* Use of a dressing or bandage covering the rash that cannot reasonably be removed for required study activities without compromising patient comfort or care.
* Patients who are pregnant will not be excluded from the study unless they present with a rash or other skin conditions that may confound assessments
* A medical condition that, in the opinion of the investigator, precludes the patient from being able to provide informed consent OR presents confounds which may bias the study outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
GLOB-IAD Clinical Assessment | 14 days
  The GLOB-IAD Clinical Assessment is the only validated clinical tool for assessing MASD. This assessment will be performed daily for the first 7 days, and once again at day 14. All GLOB-IAD assessments will be done by a qualified study team member (i.e., principle investigator, wound care nurse, etc.).
Visual Analog Scale for Erythema | 14 Days
  The Visual Analog Scale (VAS) for erythema is a visual assessment tool to measure the severity of a patient's erythema. The VAS Erythema employs a visual scale from 0 "no visible signs of erythema" to 100 "worst possible erythema", allowing the investigator to capture erythema for all skin colors and types. The VAS Erythema will be performed at baseline, day 7, and day 14.

SECONDARY OUTCOMES:
Safety - Adverse Events and Product-Related Adverse Effects | 14 Days
  Safety of the investigational product will be assessed by documenting the frequency and severity of adverse events, and their relationship to the investigational product.
Patient-reported Satisfaction | 14 Days
  On the last visit of the study, patients will be asked to fill out a questionnaire on their satisfaction with the cream used and their opinion on how effective it was at relieving symptoms and treating their rash. The satisfaction questionnaire consists of 4 sections; experience in the trial, satisfaction with the product, comparison to other products, and open feedback.
Visual Analog Scale - Symptoms | 14 Days
  The Visual Analog Scale (VAS) for symptoms is a visual assessment tool to measure the severity of a patient's symptoms of pain, itching and burning. The VAS Erythema employs a visual scale from 0 "no feelings of symptom" to 100 "worst possible symptom", allowing a nominal value to be assigned. Three VAS questions will be performed daily - for pain, burning and itching of the rash - for the duration of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calgary Cumming School of Medicine, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No